CLINICAL TRIAL: NCT04131114
Title: Suspected Glaucoma and Glaucoma After Congenital and Infantile Cataract Surgery: A Longitudinal Study in China
Brief Title: Glaucoma After Congenital And Infantile Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: CCPMOH2016-China-0303
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Glaucoma; Congenital Cataract
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pediatric patients who have undergone surgery for congenital or infantile cataracts have a risk of developing suspected glaucoma and glaucoma, but the current evidence does not address our understanding of the incidence and associated risk factors of suspected glaucoma/glaucoma for application in clinical standard care. Therefore, this study investigated the incidence of and risk factors for suspected glaucoma/glaucoma in patients who have undergone surgery for congenital/infantile cataracts.

DETAILED DESCRIPTION:
A prospective longitudinal cohort study of pediatric patients who underwent surgery for congenital/infantile cataracts between January 2011 and December 2021 was performed.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of congenital/infantile cataracts without any surgical intervention;
* age younger than 10 years;
* cataract surgery performed at the Zhongshan Ophthalmic Center after enrollment

Exclusion Criteria:

* a preoperative IOP above 21 mm Hg;
* the presence of any preoperative sign of glaucoma, such as corneal enlargement, corneal clouding, excessive optic nerve cupping, or a family history of glaucoma;
* the presence of ocular trauma or other abnormalities, such as microcornea, microphthalmia, persistent hyperplastic primary vitreous, Peters anomaly, congenital aniridia, Marfan syndrome, lens dislocation, retinitis pigmentosa, high myopia, fundus lesions, rubella, and Lowe syndrome.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A prospective longitudinal cohort study of pediatric patients who underwent surgery for congenital/infantile cataracts between January 2011 and December 2016 was performed.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of suspected glaucoma/glaucoma after congenital cataracts | 3 years
  A Kaplan-Meier analysis was used.
Risk Factors of suspected glaucoma/glaucoma after congenital cataracts | 3 years
  Cox regression analysis was assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No